CLINICAL TRIAL: NCT02860156
Title: Characterizing HIV-related Diastolic Dysfunction: A Cross Sectional Study Leveraging the NHLBI Heart Failure Clinical Research Network
Brief Title: Characterizing HIV-related Diastolic Dysfunction
Acronym: HFN_HIV
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00074493
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure; HIV; Diastolic Dysfunction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- HIV+/DD+: Subjects are HIV positive and have diastolic dysfunction
- HIV+/DD-: Subjects are HIV positive and do not have diastolic dysfunction
- HIV-/DD+: Subjects do not have HIV and have diastolic dysfunction

SUMMARY:
This is a multicenter clinical trial of a cross section of HIV+ patients with and without diastolic dysfunction. Approximately 200 HAART-treated virally suppressed HIV+ subjects (100 HIV+/DD+ & 100 HIV+/DD-) will be enrolled. This study will evaluate biomarkers, phenomapping, metabolomics, cMRI, echocardiography to determine characteristics unique to this patient population.

DETAILED DESCRIPTION:
With the advent of highly active antiretroviral therapy (HAART), human immuno¬deficiency virus (HIV) type 1 infection has become a chronic disease. The proportion of patients expected to survive 5, 10, and 15 years after conversion in the HAART era are 99%, 93% and 89% respectively. With increased life expectancy and decreased morbidity from opportunistic infections, the importance of chronic complications associated with HIV-1 infection, including HF is becoming more evident. The advent of HAART has altered the epidemiology of HIV associated cardiomyopathy evolving from a primarily left ventricular systolic dysfunction to the growing recognition of left ventricular DD. DD is associated with the development of atrial fibrillation and heart failure (HF), and portends higher risk for all-cause mortality. Thus there is a widespread prevalence of cardiac abnormalities in HIV infected individuals that are associated with HF development and may represent a sub-clinical abnormality that may be potentially intervened upon to reduce the risk of subsequent HF. There are little data to understand the natural history and pathogenesis of cardiac abnormalities, specifically DD in HIV+ individuals, which may adversely affect the longevity and quality of life of these individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Age >40 years
2. Willingness and ability to provide informed consent
3. HIV antibody positive
4. On HAART for >6 months (HIV positive cohort only)
5. History of adequate viral suppression as defined by HIV RNA level <200 copies/mL in the past 6 months
6. LVEF >50% -

Exclusion Criteria:

1. Past EF <50%
2. Moderate or severe valve stenosis or regurgitation, or past repair or replacement
3. Percutaneous or surgical revascularization or active angina
4. Persistent atrial fibrillation
5. BP>160mmHg SBP or >100mmHg DBP
6. Comorbid inflammatory disease (e.g. RA or SLE)
7. Active cancer or cancer chemotherapy treatment in the prior year (except skin cancer that did not require chemotherapy or radiation)
8. Chronic use of steroids or anti-inflammatory therapy
9. GFR <30 mL/min
10. Active in a clinical trial with investigational product
11. Pregnant or lactating females
12. Contraindication to cMR or gadolinium injection (such as severe claustrophobia, metal implants, etc.)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are receiving care at a site participating in the Heart Failure Clinical Research Network program, are HIV positive, have been on HAART for >6 months and are virally suppressed will be screened for participation.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
persistent inflammation between HIV+/DD- and HIV+/DD+ subjects | baseline visit
  Compare inflammation between HIV+/DD- and HIV+/DD+ subjects.
immune activation between HIV+/DD- and HIV+/DD+ subjects | baseline visit
  Compare immune activation between HIV+/DD- and HIV+/DD+ subjects.
inflammation between HIV+/DD- and HIV+/DD+ subjects | baseline visit
  To compare inflammation between HIV+/DD- and HIV+/DD+
Perform phenomics of aggregate demographic data to define risk factor phenotype signatures and relate these to HIV+/DD- and HIV+/DD+ subjects | baseline visit
myocardial fibrosis by magnetic resonance imaging between HIV+/DD- and HIV+/DD+ | baseline visit
  To compare myocardial fibrosis by magnetic resonance imaging between HIV+/DD- and HIV+/DD+
serum levels of biomarkers | baseline visit
  To identify systemic determinants (biomarkers) of DD in HIV+ persons
novel mechanisms underlying DD in HIV+ subjects as measured by proteomic and metabolomics panels | baseline visit
  To study the proteomic and metabolomics panels to enable identification of novel mechanisms underlying DD in HIV+ subjects
the effect of DD on mechanics of the left atrium in HIV | baseline visit
  To study the effect of DD on mechanics using left atrial strain during passive leg raise
sub-clinical necrosis in HIV+/DD+ subjects | baseline visit
  To study the sub-clinical necrosis using Troponin levels in HIV+/DD+ subjects
myocardial stress in HIV+/DD+ subjects | baseline visit
  To study myocardial stress using NTProBNP levels in HIV+/DD+ subjects
Perform phenomics of aggregate clinical data to define risk factor phenotype signatures and relate these to HIV+/DD- and HIV+/DD+ subjects | baseline visit
  Clinical data
Perform phenomics of aggregate biomarker data to define risk factor phenotype signatures and relate these to HIV+/DD- and HIV+/DD+ subjects | baseline visit
  Biomarker data
Perform phenomics of aggregate electrocardiogram data to define risk factor phenotype signatures and relate these to HIV+/DD- and HIV+/DD+ subjects | baseline visit
  electrocardiogram data
Perform phenomics of aggregate imaging data to define risk factor phenotype signatures and relate these to HIV+/DD- and HIV+/DD+ subjects | baseline visit
  imaging data

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Anstrom, PhD, Principal Investigator — Duke University Health Services; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (12):
- United States (12):
  - The Emory Clinic, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital-Washington University Hospital, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - The University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colaco NA, Wang TS, Ma Y, Scherzer R, Ilkayeva OR, Desvigne-Nickens P, Braunwald E, Hernandez AF, Butler J, Shah SH, Shah SJ, Hsue PY. Transmethylamine-N-Oxide Is Associated With Diffuse Cardiac Fibrosis in People Living With HIV. J Am Heart Assoc. 2021 Aug 17;10(16):e020499. doi: 10.1161/JAHA.120.020499. Epub 2021 Aug 7. PMID 34365799